CLINICAL TRIAL: NCT03213340
Title: A Pilot Study to Explore the Acute Effects of Phytonutrients Upon Muscle Microvascular Blood Flow (Perfusion) in Response to Feeding in Older Adults.
Brief Title: Effects of Phytonutrients Upon Muscle Perfusion in Response to Feeding
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: BL31
Record Dates: First submitted 2017-06-26; First posted 2017-07-11 (Actual); Last update posted 2020-01-31 (Actual); Status verified 2020-01

CONDITIONS: Biological Aging

STUDY DESIGN:
Intervention Model Description: 3 cohorts, crossover within cohort
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Catechin Cohort 1 (Experimental): 2 treatment - Experimental Catechin Blend; Control 1 Placebo
  Interventions: Other: Catechin Cohort 1
- Curcuminoid Cohort 2 (Experimental): 2 treatment - Experimental Curcuminoid Blend; Control 1 Placebo
  Interventions: Other: Curcuminoid Cohort 2
- Flavonoid Cohort 3 (Experimental): 2 treatment - Experimental Flavonoid Blend; Control 2 Low-Flavonoid Blend
  Interventions: Other: Flavonoid Cohort 3

INTERVENTIONS:
Other: Catechin Cohort 1 — - 4 capsules taken with water 1 hour prior to meal
  Arms: Catechin Cohort 1
Other: Curcuminoid Cohort 2 — - 2 capsules taken with water 1 hour prior to meal
  Arms: Curcuminoid Cohort 2
Other: Flavonoid Cohort 3 — - ~ 1 oz. serving consumed 30 minutes before meal
  Arms: Flavonoid Cohort 3

SUMMARY:
This is a random order cross over design trial to evaluate the efficacy of select nutritional ingredients on enhancing muscle perfusion in response to an acute meal stimulus.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) 18-30 kg/m2
* Free from active metabolic disease
* Normotensive

Exclusion Criteria:

* Habitual gym use or formal exercise (more than once a week) or other routine strenuous physical activity
* Smokers
* Surgery within past 3 months
* Active cardiovascular disease
* Taking beta-adrenergic blocking agents
* Cerebrovascular disease:
* Active respiratory disease
* Active metabolic disease
* Active inflammatory bowel or renal disease
* Active Malignancy or until confirmed remission
* Clotting dysfunction
* History of DVT
* Significant musculoskeletal or neurological disorders
* Family history of early (<55y) death from cardiovascular disease
* Known sensitivity to Sonovue contrast agent
* Known allergy or intolerance to any of the study ingredients
* Current use of any of the study ingredients

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 39 (Actual)
Dates: Start 2017-09-14 (Actual); Primary Completion 2019-10-02 (Actual); Study Completion 2019-10-02 (Actual)

PRIMARY OUTCOMES:
muscle microvascular blood flow | Baseline to 240 minutes
  contrast enhanced ultrasound

SECONDARY OUTCOMES:
muscle macrovascular blood flow | Baseline to 240 minutes
  doppler ultrasound
central vascular blood flow | Baseline to 90 minutes
  echocardiography
cerebral blood flow | Baseline to 120 minutes
  doppler ultrasound
endothelial function | Baseline to 120 minutes
  flow mediated dilation

CONTACTS AND LOCATIONS:
Overall Officials: Suzette Pereira, PhD, Study Chair — Abbott Nutrition
Locations (1):
- University of Nottingham, Derby, United Kingdom

IPD SHARING:
Plan to Share IPD: No